CLINICAL TRIAL: NCT00813644
Title: A Study of Flexible Ureteroscopy Proficiency After Training on the Uromentor Simulator
Acronym: UROSIMULATOR08
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Golan Shay, MD, Urology department, Rabin medical center
Other Study IDs: 5166
Record Dates: First submitted 2008-12-21; First posted 2008-12-23 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Endoscopic Skills

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: uromentor training
- 2: non uromentor training

SUMMARY:
The development of virtual reality (VR) simulators is changing surgical endoscopic education. The translation of VR skills into clinical endoscopic proficiency has been shown by M.PEARLE. The improvement in performing endoscopic tasks after VR training was evaluated on a cadaver. Our goal is to evaluate the performance of novice endoscopists at the operating room by a randomized controlled study comparing subjects randomized to train on a the "UroMentor" simulator to those without VR training.

ELIGIBILITY:
Inclusion Criteria:

* novice urologists without endo-urological experience

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: urologists
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-12

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Beilinson hospital, Petah Tikva, Israel